CLINICAL TRIAL: NCT05169320
Title: Patient-TAILORed Ablation of Atrial Fibrillation Drivers in Persistent Stages Based on Instantaneous Amplitude and Frequency Modulation Criteria (TAILOR-AF)
Brief Title: Patient-TAILORed Ablation of Persistent AF Guided by Instantaneous Amplitude and Frequency Modulation Maps (TAILOR-AF)
Acronym: TAILOR-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Responsible Party: Principal Investigator, David Filgueiras-Rama, Principal Investigator, Hospital San Carlos, Madrid
Other Study IDs: TAILOR-AF
Record Dates: First submitted 2021-11-26; First posted 2021-12-23 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case group: Patients with symptomatic persistent AF episodes after previous failure of ≥2 pulmonary vein isolation procedures
  Interventions: Device: Subcutaneous implantable loop recorder (ILR) implantation; Procedure: Mapping and catheter ablation; Procedure: Minimally invasive surgical ablation via thoracoscopy

INTERVENTIONS:
Device: Subcutaneous implantable loop recorder (ILR) implantation — All patients will undergo subcutaneous implantable loop recorder (ILR) implantation to quantify AF burden 1 month before the ablation procedure and at least 1 year after the ablation procedure.
Procedure: Mapping and catheter ablation — Driver regions will be identified during persistent AF using a conventional electroanatomical mapping system, multielectrode mapping catheters, and leading-driver maps generated by novel single-signal algorithms based on an automatic and accurate analysis of the instantaneous amplitude and frequency modulations displayed by atrial signals (iAM and iFM, respectively). Such maps enable the location of the spatiotemporally stable regions that drive persistent AF (leading drivers). Leading-driver regions that can be reasonably targeted/isolated with catheter ablation without high-risk of complications upon radiofrequency delivery will be targeted for ablation.
Procedure: Minimally invasive surgical ablation via thoracoscopy — This procedure will be performed only in those patients whose leading-driver maps in the previous mapping and catheter ablation procedure fulfill the following requirements:
  1. Extensive atrial remodeling who will not likely get any benefit from catheter-based ablation due to too large atrial leading driver areas (≥10-15% of atrial surface), or
  2. Leading drivers located at regions with high-risk of complications upon radiofrequency delivery (e.g. left and right atrial appendages, coronary sinus, in the vicinity [≤5 mm] of the cardiac specific conduction system).
  In such patients, the leading-driver regions not completely targeted or not targeted at all in the previous index mapping and catheter ablation procedure, will be specifically ablated/isolated by minimally invasive surgical ablation techniques via thoracoscopy.

SUMMARY:
Pulmonary vein isolation (PVI) is still considered the cornerstone of catheter ablation for patients with persistent atrial fibrillation (AF). However, ablation outcomes in patients with persistent AF are suboptimal with high recurrence rates after a single PVI procedure.

Recently, the investigators developed a new strategy, which enables precise identification of the driver regions allegedly responsible for the maintenance of persistent AF outside the pulmonary veins. This approach uses a conventional electroanatomical mapping system and novel single-signal algorithms based on automatic and accurate analysis of the instantaneous amplitude and frequency modulations displayed by atrial signals during AF (iAM and iFM, respectively) to locate the spatiotemporally stable regions that drive persistent AF (leading drivers).

This strategy also enables to identify highly complex substrates in which targeting leading driver regions with catheter-based ablation may not be feasible or could be potentially associated with a significantly higher risk of complications. In such patients, the iAM/iFM maps obtained in the index catheter mapping and ablation procedure will be used to guide an additional patient-specific, minimally invasive surgical ablation approach via thoracoscopy, aiming to completely but specifically target all leading driver regions.

The main objective of the TAILOR-AF study is to identify (via iAM/iFM maps), target and ablate AF leading drivers in patients with symptomatic persistent AF recurrences despite ≥2 previous PVI procedures. The methods include a percutaneous catheter mapping and ablation approach followed by a minimally invasive surgical approach via thoracoscopy, if necessary. As a secondary objective we will study the association of underlying blood biomarkers, atrial imaging and surface ECG parameters, with advanced remodeling stages requiring a surgical approach to target leading driver regions.

This is a single center study (Hospital Clínico San Carlos, Madrid, Spain) that will recruit 25 patients with symptomatic persistent AF episodes despite having been submitted to ≥2 PVI prior procedures. All patients will undergo subcutaneous implantable loop recorder (ILR) implantation to address AF burden 1 month before the ablation procedure and at least 1 year after the ablation procedure. The primary outcome of the study will be AF freedom after one year of follow-up off antiarrhythmic drugs.

DETAILED DESCRIPTION:
The study is co-sponsored by the Fundación para la Investigación Biomédica del Hospital Clínico San Carlos (Madrid, Spain) and the Centro Nacional de Investigaciones Cardiovasculares Carlos III (F.S.P.) (Madrid, Spain).

Dr. David Filgueiras-Rama (MD, PhD, affiliation: Hospital Clínico San Carlos) and Dr. Jorge G. Quintanilla (MScEng, PhD, affiliation: Centro Nacional de Investigaciones Cardiovasculares [CNIC]) are Co-Principal Investigators of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic persistent AF (defined as a sustained episode lasting ≥ 7 days) despite ≥2 previous PVI, with or without other atrial anatomical targets isolated in previous procedures (e.g. superior vena cava, coronary sinus or others).
2. AF episodes refractory to ≥1 antiarrhythmic drug (flecainide, propofenone, amiodarone or droneradore) or adverse events related to antiarrhythmic drugs that do not allow long-term drug therapy.
3. Age between 18-75 years old.
4. Patients must be willing and able to comply with all peri-ablation and follow-up requirements.
5. Signed informed consent.
6. Confirmed pulmonary vein isolation in the index (in current protocol) procedure.

Exclusion Criteria:

1. Patients with paroxysmal AF (defined as a sustained episode lasting < 7 days).
2. Patients for whom cardioversion or sinus rhythm will never be attempted/pursued.
3. Patients with AF secondary to an obvious reversible cause.
4. Patients with contraindications to systemic anticoagulation with heparin or coumadin or a direct thrombin inhibitor.
5. Non-sustained AF during the mapping procedure.
6. Severe underlying systemic disease (e.g. dementia, any end-disease stage, sepsis, etc).
7. Severe left atrial dilation (left atrial volume >73 ml/m2).
8. Severe underlying cardiac disease (e.g. left ventricular ejection fraction ≤35%, severe non-corrected valvular disease, severe non-corrected coronary artery disease, hypertrophic cardiomyopathy, other inherited arrhythmia syndromes, severe dilated cardiomyopathy with NYHA functional class III, IV).
9. Hemodynamic instability due to any cardiac or non-cardiac disease.
10. Pregnancy.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from the Cardiored1 program (including 4 hospitals in Madrid, Spain) with symptomatic persistent AF in spite of ≥2 PVI previous procedures.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Fibrillation without antiarrhythmic drugs | After one year of follow-up
  Number/Percentage of participants with freedom from Atrial Fibrillation without antiarrhythmic drugs

SECONDARY OUTCOMES:
Acute termination of Atrial Fibrillation during the procedure/s | During catheter ablation and/or minimally invasive thoracoscopic surgical procedures
  Number/Percentage of participants with acute termination of Atrial Fibrillation during the procedure/s
Freedom from Atrial Fibrillation with or without antiarrhythmic drugs | After one year of follow-up
  Number/Percentage of participants with freedom from Atrial Fibrillation with or without antiarrhythmic drugs
Freedom from Atrial Tachycardia/Flutter with or without antiarrhythmic drugs | After one year of follow-up
  Number/Percentage of participants with freedom from Atrial Tachycardia/Flutter with or without antiarrhythmic drugs

OTHER OUTCOMES:
Comparison of pre-ablation dominant frequencies in atrial electrocardiogram in Hz between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-ablation dominant frequencies in atrial electrocardiogram in Hz (after QRST subtraction) will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up
Comparison of pre-ablation coefficients of variation of dominant frequencies in 12-lead atrial electrocardiogram (Hz/Hz), between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-ablation coefficients of variation (median/interquartile range, Hz/Hz) of dominant frequencies in 12-lead atrial electrocardiogram, will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of the relative difference (%) of intra-procedure pre-ablation and post-ablation dominant frequencies in atrial electrocardiogram, between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  The relative difference of intra-procedure pre-ablation and post-ablation dominant frequencies in atrial electrocardiogram after QRST subtraction ([DFpost-DFpre]*100/DFpre) will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up. If electrical cardioversion is performed intraprocedurally to restore sinus rhythm after ablation, the post-ablation measurements will be performed after completion of ablation and prior to electrical cardioversion.
Comparison of ratio (adimensional) of intra-procedure pre-ablation and post-ablation coefficients of variation of dominant frequencies in 12-lead atrial electrocardiogram, between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Ratio (adimensional) between intra-procedure pre-ablation and post-ablation coefficients of variation (median/interquartile range) of dominant frequencies in 12-lead atrial electrocardiogram after QRST subtraction, will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.If electrical cardioversion is performed intraprocedurally to restore sinus rhythm after ablation, the post-ablation measurements will be performed after completion of ablation and prior to electrical cardioversion.
Comparison of pre-procedure values of Galectin-3 (ng/mL) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure samples of peripheral blood will be collected in all patients. Galectin-3 values (ng/mL) from these samples will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of pre-procedure values of Interleukin1-ß (pg/mL) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure samples of peripheral blood will be collected in all patients. Interleukin1-ß values (pg/mL) from these samples will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of pre-procedure values of Tumor Necrosis Factor-α (pg/mL) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure samples of peripheral blood will be collected in all patients. Tumor necrosis factor-α values (pg/mL) from these samples will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of pre-procedure values of Interleukin-6 (pg/mL) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure samples of peripheral blood will be collected in all patients. Interleukin-6 (pg/mL) from these samples will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of pre-procedure values of procollagen III terminal propeptide (pg/mL) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure samples of peripheral blood will be collected in all patients. Procollagen III terminal propeptide (pg/mL) from these samples will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of pre-procedure values of procollagen I terminal propeptide (ng/mL) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure samples of peripheral blood will be collected in all patients. Procollagen I terminal propeptide (ng/mL) from these samples will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of pre-procedure values of cross linked C terminal telopeptide of type I collagen (ng/mL) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure samples of peripheral blood will be collected in all patients. Procollagen I terminal propeptide (ng/mL) from these samples will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of pre-procedure values of echocardiography-based rigth atrium area (mm2) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure echocardiographic imaging will be performed in all patients. Right atrium area (mm2) will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of pre-procedure values of echocardiography-based left atrium area (mm2) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure echocardiographic imaging will be performed in all patients. Left atrium area (mm2) will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.
Comparison of pre-procedure values of echocardiographic/computational tomography 3-dimensional left atrium volume index (mL/m2) between patients with and without Atrial Fibrillation recurrence | After one year of follow-up
  Pre-procedure echocardiographic/computational tomography imaging will be performed in all patients. 3-dimensional left atrium volume index (mL/m2) will be compared between patients with and without Atrial Fibrillation recurrence after one year of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: David Filgueiras-Rama, MD, PhD, Principal Investigator — Hospital Clínico San Carlos & CNIC
Locations (2):
- Spain (2):
  - Centro Nacional de Investigaciones Cardiovasculares (CNIC), Madrid
  - Hospital Clínico San Carlos, Madrid

REFERENCES:
- [Background] Quintanilla JG, Alfonso-Almazan JM, Perez-Castellano N, Pandit SV, Jalife J, Perez-Villacastin J, Filgueiras-Rama D. Instantaneous Amplitude and Frequency Modulations Detect the Footprint of Rotational Activity and Reveal Stable Driver Regions as Targets for Persistent Atrial Fibrillation Ablation. Circ Res. 2019 Aug 30;125(6):609-627. doi: 10.1161/CIRCRESAHA.119.314930. Epub 2019 Aug 1. PMID 31366278
- [Background] Rosa G, Quintanilla JG, Salgado R, Gonzalez-Ferrer JJ, Canadas-Godoy V, Perez-Villacastin J, Perez-Castellano N, Jalife J, Filgueiras-Rama D. Mapping Technologies for Catheter Ablation of Atrial Fibrillation Beyond Pulmonary Vein Isolation. Eur Cardiol. 2021 May 17;16:e21. doi: 10.15420/ecr.2020.39. eCollection 2021 Feb. PMID 34093742
- [Background] Quintanilla JG, Shpun S, Jalife J, Filgueiras-Rama D. Novel approaches to mechanism-based atrial fibrillation ablation. Cardiovasc Res. 2021 Jun 16;117(7):1662-1681. doi: 10.1093/cvr/cvab108. PMID 33744913
- See also: Eur Cardiol. 2021 May 17;16:e21. — https://www.ecrjournal.com/articles/mapping-technologies-catheter-ablation-atrial-fibrillation-beyond-pulmonary-vein-isolation